CLINICAL TRIAL: NCT04777201
Title: A Multicenter, Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of Faricimab in Patients With Neovascular Age-Related Macular Degeneration (AVONELLE-X)
Brief Title: A Study to Evaluate the Long-Term Safety and Tolerability of Faricimab in Participants With Neovascular Age-Related Macular Degeneration
Acronym: AVONELLE-X
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GR42691; 2020-004523-16 (EudraCT Number)
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — faricimab

STUDY DESIGN:
Masking Description: The first 12 weeks of the main study will be a masked period (to transition from the multi-arm parent studies) during which participants may receive either faricimab or sham injection. Participants and physicians will be masked only to the faricimab treatment interval. After the Week 12 treatment procedure, this study will follow an open-label design. The BCVA examiner will remain masked for the duration of the main long-term extension study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Main Study: Faricimab PTI (Experimental)
  Interventions: Drug: Faricimab; Other: Sham Procedure; Drug: Anti-VEGF Therapy
- Substudy: Faricimab PTI (Experimental)
  Interventions: Drug: Faricimab; Drug: Anti-VEGF Therapy

INTERVENTIONS:
Drug: Faricimab — Faricimab 6 mg will be administered by intravitreal (IVT) injection into the study eye according to the personalized treatment interval (PTI) dosing regimen for the duration of the study.
  Other Names: RO6867461; RG7716
Other: Sham Procedure — The sham is a procedure that mimics an IVT injection and involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. The sham procedure will be administered to participants as appropriate during the first 12 weeks of this study in order to maintain the masking of the initial faricimab PTI.
  Arms: Main Study: Faricimab PTI
Drug: Anti-VEGF Therapy — At the discretion of the principal investigator, participants were allowed to have their fellow (non-study) eye treated with the standard of care anti-VEGF therapy (if needed) according to region-specific anti-VEGF prescribing information for the recommended dose and frequency of treatment.

SUMMARY:
This main long-term extension study is designed to evaluate the long-term safety and tolerability of faricimab 6 milligrams (mg) administered by intravitreal injection at a personalized treatment interval (PTI) to participants with neovascular age-related macular degeneration (nAMD) who enrolled in and completed one of the Phase III studies: GR40306 (NCT03823287) or GR40844 (NCT03823300), also referred to as the parent studies. Eligible patients who consent to participate in this main study will be enrolled upon completion of the end-of-study visit in the parent study.

Additionally, there is a substudy that is being conducted. The aim of this substudy is to evaluate the impact of intravitreal faricimab on the health of the corneal endothelial cells in the study eyes of patients with nAMD to fulfill a U.S. Food and Drug Administration (FDA) post-marketing requirement. The fellow eyes of the same enrolled participants in the substudy will serve as the controls.

ELIGIBILITY:
Inclusion Criteria for the Main Study:

* Previous enrollment in and completion of Study GR40306 (NCT03823287) or Study GR40844 (NCT03823300), without study or study drug discontinuation
* For women of childbearing potential: agreement to remain abstinent or use contraception, and agreement to refrain from donating eggs. Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 3 months after the final dose of faricimab. Women must refrain from donating eggs during the same period.

Inclusion Criteria for the Substudy:

* In addition to all inclusion criteria specified in the main Study GR42691, participants in the Substudy must meet the following criteria:
* Sign an informed consent form for the Substudy
* Must be able to participate for at least 48 weeks in the Substudy and have at least the first visit while enrolled in the main Study GR42691
* A difference of <10% in corneal endothelial cell density at screening between the two eyes as measured by specular microscopy and determined by the independent reading center

Exclusion Criteria for the Main Study:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of faricimab
* Presence of other ocular diseases that give reasonable suspicion of a disease or condition that contraindicates the use of faricimab, that might affect interpretation of the results of the study or that renders the patient at high risk for treatment complications
* Presence of other diseases, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of faricimab and that might affect interpretation of the results of the study or that renders the patient at high risk of treatment complications
* History of a severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the faricimab injections, study-related procedure preparations, dilating drops, or any of the anesthetic and antimicrobial preparations used by a patient during the study
* Requirement for continuous use of any medications or treatments indicated as prohibited therapy

Exclusion Criteria for the Substudy:

In addition to the exclusion criteria specified in the main Study GR42691, patients will be excluded from this substudy if they meet any of the following exclusion criteria:

* Prior and/or current administration of faricimab in the fellow (non-study) eye
* Prior administration of brolucizumab in the fellow (non-study) eye

Exclusion Criteria in Either Eye for the Substudy:

* Corneal endothelial cell density ≤1500 cells/mm2 in either eye at screening as determined by the independent corneal reading center
* Fuchs endothelial corneal dystrophy Grade ≥2
* Previous ocular trauma (blunt or penetrating) and/or corneal endothelial cell damage, including from blunt or surgical trauma (including complicated cataract surgery resulting in complicated lens placement such as anterior chamber intraocular lens, sulcus intraocular lens, aphakia, etc.)
* Any ocular condition that precludes obtaining an analyzable specular microscopy image
* Active or history of corneal edema
* Any active or history of corneal dystrophies, excluding Fuchs endothelial corneal dystrophy Grade <2
* Active or history of iridocorneal endothelial syndrome
* Active or history of pseudoexfoliation syndrome
* Active or history of herpetic keratitis or kerato-uveitis (including herpes simplex virus and herpes zoster virus)
* Intraocular laser therapy including selective laser trabeculoplasty, yttrium-aluminum garnet (YAG), prophylactic peripheral iridotomy within 1 year of screening, or YAG capsulotomy within 3 months of screening
* Prior vitrectomy surgery, submacular surgery, or other surgical intervention for AMD
* Prior pars plana vitrectomy surgery
* Previous intraocular device implantation excluding intraocular lenses
* Cataract surgery within 6 months of screening or planned for during the study
* History of glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery. Other types of prior glaucoma surgery are allowed providing that the surgery occur more than 6 months before screening
* Administration of topical Rho kinase inhibitors (e.g., Rhopressa eye drops) within 1 month prior to the screening visit
* Contact lens wear in either eye within 2 months of screening
* History of corneal transplantation, including partial-thickness corneal grafts (e.g., Descemet membrane endothelial keratoplasty, Descemet stripping endothelial keratoplasty)
* Active or history of iridocorneal endothelial syndrome
* Active or history of pseudoexfoliation syndrome

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1036 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (251):
- United States (85):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - Retinal Diagnostic Center, Campbell, California
  - The Retina Partners, Encino, California
  - South Coast Retina Center, Los Angeles, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Southern CA Desert Retina Cons, Palm Desert, California
  - California Eye Specialists Medical group Inc., Pasadena, California
  - Retina Consultants, San Diego, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - University of California, Davis, Eye Center, Sacramento, California
  - Retinal Consultants Med Group, Sacramento, California
  - Orange County Retina Med Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Retina Consultants of Southern, Colorado Springs, Colorado
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Rand Eye, Deerfield Beach, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Northwestern Medical Group/Northwestern University, Chicago, Illinois
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Prairie Retina Center, Springfield, Illinois
  - Raj K. Maturi, MD PC, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, Lenexa, Kansas
  - Maine Eye Center, Portland, Maine
  - Retina Specialists, Baltimore, Maryland
  - The Retina Care Center, Baltimore, Maryland
  - Johns Hopkins Med, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - VitreoRetinal Surgery, PLLC., Edina, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Retina Associates of St. Louis, Florissant, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Mid Atlantic Retina - Wills Eye Hospital, Cherry Hill, New Jersey
  - NJ Retina, Edison, New Jersey
  - Retina Associates of NJ, Teaneck, New Jersey
  - Long Is. Vitreoretinal Consult, Great Neck, New York
  - Ophthalmic Cons of Long Island, Oceanside, New York
  - Retina Assoc of Western NY, Rochester, New York
  - Vitreoretinal Consultants of New York, Shirley, New York
  - The Retina Consultants, Slingerlands, New York
  - Retina Vit Surgeons/Central NY, Syracuse, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Graystone Eye, Winston-Salem, North Carolina
  - Cincinnati Eye Institute, Blue Ash, Ohio
  - Retina Assoc of Cleveland Inc, Cleveland, Ohio
  - The Ohio State University Havener Eye Institute, Columbus, Ohio
  - Midwest Retina, Dublin, Ohio
  - Retina Northwest, Portland, Oregon
  - Charleston Neuroscience Inst, Ladson, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates Chattanooga, Chattanooga, Tennessee
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC., Nashville, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Texas, Houston, Texas
  - Valley Retina Institute P.A., McAllen, Texas
  - Retina Center of Texas, Southlake, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, PLLC, Salt Lake City, Utah
  - Rocky Mountain Retina, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Institute, Norfolk, Virginia
  - Pacific Northwest Retina, Silverdale, Washington
- Argentina (7):
  - Organizacion Medica de Investigacion, Buenos Aires
  - Fundacion Zambrano, CABA
  - Centro Oftalmologico Dr. Charles S.A., Capital Federal
  - Oftalmos, Capital Federal
  - Buenos Aires Mácula, Ciudad Autonoma Buenos Aires
  - Oftar, Mendoza
  - Grupo Laser Vision, Rosario
- Australia (7):
  - Eyeclinic Albury Wodonga, Albury, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Sydney West Retina, Westmead, New South Wales
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- Austria (2):
  - LKH-Univ.Klinikum Graz, Graz
  - Medizinische Universitat Wien, Vienna
- Brazil (2):
  - Hospital de Olhos de Aparecida - HOA, Aparecida de Goiânia, Goiás
  - Universidade Federal de Sao Paulo - UNIFESPX, São Paulo, São Paulo
- Bulgaria (2):
  - Pentagram Eye Hospital (Medical Center "Pentagram"), Sofia
  - Specialized Hospital for Active Treatment of Eye Diseases Zora, Sofia
- Canada (7):
  - Calgary Retina Consultants, Calgary, Alberta
  - University of British Columbia - Vancouver Coastal Health Authority, Vancouver, British Columbia
  - Ivey Eye Institute, London, Ontario
  - Retina Institute of Ottawa, Ottawa, Ontario
  - Toronto Retina Institute, Toronto, Ontario
  - Institut De L'Oeil Des Laurentides, Boisbriand, Quebec
  - Michel Giunta Clinique Medical, Sherbrooke, Quebec
- Denmark (2):
  - Rigshospitalet Glostrup, Glostrup Municipality
  - Sjællands Universitetshospital, Roskilde, Roskilde
- France (6):
  - Chi De Creteil, Créteil
  - Pole Vision Val d'Ouest, Écully
  - Hopital de la croix rousse, Lyon
  - Centre Paradis Monticelli, Marseille
  - CHU Nantes - Hotel Dieu, Nantes
  - Hopital Lariboisiere, Paris
- Germany (6):
  - Universitatsklinikum Koln, Cologne
  - Universitätkslinikum Düsseldorf, Augenklinik, Düsseldorf
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Universitätsklinik Heidelberg, Heidelberg
  - Augenabteilung am St. Franziskus-Hospital, Münster
  - Universitatsklinikum Munster, Münster
- Hong Kong (2):
  - The University of Hong Kong, Hong Kong
  - Hong Kong Eye Hospital, Mong Kok
- Hungary (7):
  - Eszak-Pesti Centrumkorhaz - Honvedkorhaz, Budapest
  - Bajcsy-Zsilinszky Hospital, Budapest
  - Budapest Retina Associates Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecem
  - Ganglion Medial Center, Pécs
  - Szegedi Tudományegyetem ÁOK, Szeged
  - Zala Megyei Kórház, Zalaegerszeg
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah MC, Jerusalem
  - Rabin MC, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky MC, Tel Aviv
- Italy (5):
  - Fondazione G.B. Bietti Per Lo Studio E La Ricerca in Oftalmologia-Presidio Ospedaliero Britannico, Rome, Lazio
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico-Clinica Regina Elena, Milan, Lombardy
  - Asst Fatebenefratelli Sacco, Milan, Lombardy
  - Nuovo Ospedale S. Chiara - A.O.U.P Presidio Ospedaliero di Cisanello, Pisa, Tuscany
  - Azienda Ospedaliera di Perugia Ospedale S. Maria Della Misericordia, Perugia, Umbria
- Japan (36):
  - Nagoya University Hospital, Aichi
  - Nagoya City University Hospital, Aichi
  - Aichi Medical University Hospital, Aichi
  - Daiyukai Daiichi Hospital, Aichi
  - Chiba University Hospital, Chiba
  - Toho University Sakura Medical Center, Chiba
  - Hayashi Eye Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Sapporo City General Hospital, Hokkaido
  - Asahikawa Medical University Hospital, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center (Hyogo AGMC), Hyōgo
  - Hyogo Medical University Hospital, Hyōgo
  - Kozawa eye hospital and diabetes center, Ibaraki
  - Kagawa University Hospital, Kagawa
  - Kagoshima University Hospital, Kagoshima
  - Ideta Eye Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Mie University Hospital, Mie
  - Fukushima Medical University Hospital, Miyagi
  - University of Miyazaki Hospital, Miyazaki
  - Shinshu University Hospital, Nagano
  - Iida Municipal Hospital, Nagano
  - Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Nara Medical University Hospital, Nara
  - University of the Ryukyus Hospital, Okinawa
  - Kitano Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Kansai Medical University Medical Center, Osaka
  - Kansai Medical University Hospital, Osaka
  - National Defense Medical College Hospital, Saitama
  - Shiga University Of Medical Science Hospital, Shiga
  - Nihon University Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
  - Yamaguchi University Hospital, Yamaguchi
- Mexico (3):
  - Centro Oftalmológico Mira, S.C, Del. Cuauhtemoc, Mexico CITY (federal District)
  - Macula Retina Consultores, Mexico City, Mexico CITY (federal District)
  - Montemayor & Asociados (Oftalmologos), Monterrey Nuevo LEON, Nuevo León
- Het Oogziekenhuis Rotterdam, Rotterdam, Netherlands
- Poland (11):
  - Szpital sw. Lukasza, Bielsko-Biala
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Specjalistyczny O?rodek Okulistyczny Oculomedica, Bydgoszcz
  - Szpital Specjalistyczny nr 1, Bytom
  - Dobry Wzrok Sp Z O O, Gda?sk
  - Optimum Profesorskie Centrum Okulistyki, Gda?sk
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - Centrum Medyczne Dietla 19 Sp. Z O.O., Krakow
  - SP ZOZ Szpital Uniwersytecki w Krakowie Oddzia? Kliniczny Okulistyki i Onkologii Okulistycznej, Krakow
  - Caminomed, Tarnowskie Góry
  - SPEKTRUM Osrodek Okulistyki Klinicznej, Wroclaw
- Portugal (2):
  - Centro Hospitalar E Universitário de Coimbra EPE - Serviço Oftalmologia, Coimbra
  - Hospital de Sao Joao, Porto
- Russia (6):
  - Intersec Research and Technology Complex ?Eye Microsurgery? n.a. S.N. Fyodorov, Cheboksary, Mariy-El Republic
  - FSBI ?Scientific Research Institute of Eye Diseases? of Russian Academy of medical Sciences, Moscow, Moscow Oblast
  - Medical Military Academy n.a S.M.Kirov, Saint Petersburg, Sankt-Peterburg
  - 1 Saint-Petersburg St. Med. University named after academician I.P.Pavlov, Saint Petersburg, Sankt-Peterburg
  - Clinics of Eye Diseases, LLC, Kazan', Tatarstan Republic
  - ?Intersec Research and Technology Complex Eye Microsurgery n a Fyodorov Novosibirsk Branch, Novosibirsk
- Singapore Eye Research Institute, Singapore, Singapore
- South Korea (8):
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Nune Eye Hospital, Seoul
- Spain (13):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, San Cugat Del Valles, Barcelona
  - Instituto Oftalmologico Gomez Ulla, Santiago de Compostela, LA Coruna
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Instituto Oftalmologico Fernandez Vega, Oviedo, Principality of Asturias
  - Oftalvist Valencia, Burjassot, Valencia
  - Institut de la Macula i la retina, Barcelona
  - Hospital dos de maig, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Clinica Baviera, Madrid
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
- Vista Klinik Ophthalmologische Klinik, Binningen, Switzerland
- Taiwan (3):
  - Changhua Christian Hospital, Changhua
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- Turkey (Türkiye) (7):
  - Hacettepe University Medical Faculty, Ankara
  - Ankara University Medical Faculty, Ankara
  - Ankara Baskent University Medical Faculty, Ankara
  - Gazi University Faculty of Medicine, Ankara
  - Ege University Medical Faculty, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Selcuk University Faculty of Medicine, Konya
- United Kingdom (14):
  - Opthalmology Research Office, Bradford
  - Bristol Eye Hospital, Bristol
  - University Hospital of Wales, Cardiff
  - Frimley Park Hospital, Frimley
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucestershire
  - Hull Royal Infirmary, Hull
  - St James University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Manchester Royal Eye Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - New Cross Hospital, Wolverhampton
  - The York Hospital, York

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1036 participants were enrolled in the main study, 7 of whom were excluded from analysis, resulting in a final analysis set of 1029 participants. A subgroup of 117 also participated concurrently in the substudy. Only 1 eye for each participant was assigned as the study eye in the prior parent studies, per the eligibility criteria, to receive study intervention; that study eye remained the same in this main study and substudy. The fellow (other) eye was not assigned to an intervention.
Pre-assignment Details: A total of 7 patients were not included in the analysis set prior to assignment. This was a precautionary measure following a Good Clinical Practice (GCP) non-compliance audit finding at a single clinical trial site for a different investigational product.
Groups:
- Main Study Cohort A: Faricimab PTI (Prior Faricimab): This cohort included participants previously randomized to Arm A (faricimab up to every 16 weeks [Q16W]) in the parent studies [GR40306 (NCT03823287) or GR40844 (NCT03823300)]. In this long-term extension study, faricimab 6 mg was administered by intravitreal (IVT) injection into the study eye according to the personalized treatment interval (PTI) dosing regimen for the duration of the study.
- Main Study Cohort B: Faricimab PTI (Prior Aflibercept): This cohort included participants previously randomized to Arm B (aflibercept 2mg Q8W) in the parent studies [GR40306 (NCT03823287) or GR40844 (NCT03823300)]. In this long-term extension study, faricimab 6 mg was administered by intravitreal (IVT) injection into the study eye according to the personalized treatment interval (PTI) dosing regimen for the duration of the study.
- Substudy: Faricimab PTI: Participants from the main long-term extension study who also consented to participate in this substudy received faricimab 6 mg by intravitreal (IVT) injection into the study eye according to the personalized treatment interval (PTI) dosing regimen for the duration of the study. The participant's fellow eye was not assigned to an intervention. At the discretion of the principal investigator, a participant may have had their fellow eye treated with anti-VEGF therapy licensed for ocular use if the participant was diagnosed with an ocular condition for which the selected anti-VEGF therapy was approved by the country's regulatory agency. Administration of the following therapies to the fellow eye were prohibited during the substudy: faricimab, brolucizumab, bevacizumab, and Port Delivery System implantation.
Period: Main Study
Arm/Group | Main Study Cohort A: Faricimab PTI (Prior Faricimab) | Main Study Cohort B: Faricimab PTI (Prior Aflibercept) | Substudy: Faricimab PTI
Started (Participants Enrolled in Main Study) | 524 | 505 | 0
Safety-Evaluable Population (Participants Treated with Faricimab) | 520 | 505 | 0
Completed | 453 | 415 | 0
Not Completed | 71 | 90 | 0
Not completed — Withdrawal by Subject | 19 | 27 | 0
Not completed — Death | 13 | 27 | 0
Not completed — Subject missed the safety follow-up visit | 9 | 10 | 0
Not completed — Physician Decision | 8 | 10 | 0
Not completed — Adverse Event | 8 | 8 | 0
Not completed — Lost to Follow-up | 9 | 4 | 0
Not completed — Reason not specified | 3 | 3 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Substudy (Concurrent With Main Study)
Arm/Group | Main Study Cohort A: Faricimab PTI (Prior Faricimab) | Main Study Cohort B: Faricimab PTI (Prior Aflibercept) | Substudy: Faricimab PTI
Started (Participants Enrolled in the Substudy) | 0 | 0 | 117
Modified Intent-to-Treat and Safety-Evaluable Population (Participants Treated with Faricimab) | 0 | 0 | 113
Completed the Year 1 Substudy Visit (Participants Treated with Faricimab and Completed the Year 1 Visit) | 0 | 0 | 104 (99 participants completed the Year 1 visit within the analysis window (Weeks 48 to 64) and 5 completed it outside of the analysis window.)
Completed | 0 | 0 | 107 (3 of the participants completed the substudy, but they did not receive treatment with faricimab during the substudy and were excluded from analysis.)
Not Completed | 0 | 0 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Prohibited Medication | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Cataract Surgery | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The number enrolled in the GR42691 main study and overall was 1036 participants, 7 of whom were excluded from analysis as an outcome of the GCP non-compliance audit finding at one site. Therefore, 1029 participants in total were included for analysis of the main study. The GR42691 substudy enrolled a subgroup of 117 participants from the main study; 113 of those participants received at least one injection of faricimab in the study eye during the substudy and were included for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study Cohort A: Faricimab PTI (Prior Faricimab) | Main Study Cohort B: Faricimab PTI (Prior Aflibercept) | Substudy: Faricimab PTI | Total
Number analyzed (Participants) | 524 | 505 | 113 | 1142
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The GR42691 main study and substudy populations are analyzed separately. The overall number included for analysis in the main study was 1029 participants. The substudy included a subset of 113 participants who received at least one injection of faricimab in the study eye during the substudy for analysis.
  Years
    Main Study: number analyzed (Participants) | 524 | 505 | 0 | 1029
    Main Study | 76.4 (8.2) | 77.7 (8.8) |  | 77.0 (8.5)
    Substudy: number analyzed (Participants) | 0 | 0 | 113 | 113
    Substudy |  |  | 75.6 (8.1) | 75.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The GR42691 main study and substudy populations are analyzed separately. The overall number included for analysis in the main study was 1029 participants. The substudy included a subset of 113 participants who received at least one injection of faricimab in the study eye during the substudy for analysis.
  Participants
    Main Study: number analyzed (Participants) | 524 | 505 | 0 | 1029
    Main Study: Female | 308 | 291 | 0 | 599
    Main Study: Male | 216 | 214 | 0 | 430
    Substudy: number analyzed (Participants) | 0 | 0 | 113 | 113
    Substudy: Female | 0 | 0 | 61 | 61
    Substudy: Male | 0 | 0 | 52 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The GR42691 main study and substudy populations are analyzed separately. The overall number included for analysis in the main study was 1029 participants. The substudy included a subset of 113 participants who received at least one injection of faricimab in the study eye during the substudy for analysis.
  Participants
    Main Study: number analyzed (Participants) | 524 | 505 | 0 | 1029
    Main Study: Hispanic or Latino | 50 | 53 | 0 | 103
    Main Study: Not Hispanic or Latino | 463 | 445 | 0 | 908
    Main Study: Unknown or Not Reported | 11 | 7 | 0 | 18
    Substudy: number analyzed (Participants) | 0 | 0 | 113 | 113
    Substudy: Hispanic or Latino | 0 | 0 | 23 | 23
    Substudy: Not Hispanic or Latino | 0 | 0 | 90 | 90
    Substudy: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The GR42691 main study and substudy populations are analyzed separately. The overall number included for analysis in the main study was 1029 participants. The substudy included a subset of 113 participants who received at least one injection of faricimab in the study eye during the substudy for analysis.
  Participants
    Main Study: number analyzed (Participants) | 524 | 505 | 0 | 1029
    Main Study: American Indian or Alaska Native | 2 | 2 | 0 | 4
    Main Study: Asian | 76 | 83 | 0 | 159
    Main Study: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Main Study: Black or African American | 1 | 5 | 0 | 6
    Main Study: White | 433 | 402 | 0 | 835
    Main Study: More than one race | 0 | 1 | 0 | 1
    Main Study: Unknown or Not Reported | 12 | 12 | 0 | 24
    Substudy: number analyzed (Participants) | 0 | 0 | 113 | 113
    Substudy: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Substudy: Asian | 0 | 0 | 0 | 0
    Substudy: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Substudy: Black or African American | 0 | 0 | 1 | 1
    Substudy: White | 0 | 0 | 112 | 112
    Substudy: More than one race | 0 | 0 | 0 | 0
    Substudy: Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Ocular Adverse Events in the Study Eye, With Severity Determined According to Adverse Event Severity Grading Scale
Description: This is an analysis of participants with at least one ocular adverse event (AE) that occurred in the study eye. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of the seriousness, severity (e.g., mild, moderate, or severe intensity), and causality for each AE. AEs of special interest (AESI) included the following: Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, are associated with severe intraocular inflammation (IOI), or require surgical or medical intervention to prevent permanent loss of sight; suspected transmission of an infectious agent by the study drug; and, cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: From the date of first administration of faricimab through 28 days after the end of study (up to 2 years)
Population: Safety-Evaluable Population: all participants who enrolled in the long-term extension (LTE) study and received at least one dose of faricimab in the study eye during the LTE.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Cohort A: Faricimab PTI (Prior Faricimab) | Main Study Cohort B: Faricimab PTI (Prior Aflibercept) | Substudy: Faricimab PTI
Number analyzed (Participants) | 520 | 505 | 113
Participants
  Any Adverse Event (AE), Any Severity | 188 | 207 | 16
  AEs by Severity: Mild | 114 | 106 | 11
  AEs by Severity: Moderate | 58 | 75 | 4
  AEs by Severity: Severe | 13 | 23 | 1
  AEs by Severity: Missing | 3 | 3 | 0
  Serious Adverse Event (SAE) | 18 | 27 | 1
  AE Leading to Withdrawal from Study Treatment | 4 | 5 | 0
  Treatment-related AE | 8 | 12 | 2
  Treatment-related SAE | 1 | 3 | 1
  Any AE of Special Interest (AESI) | 15 | 21 | 1
  AESI: Drop in Visual Acuity Score ≥30 Letters | 11 | 16 | 1
  AESI: Associated with Severe IOI | 1 | 2 | 0
  AESI: Intervention Required to Prevent Permanent Vision Loss | 3 | 3 | 0
  AESI: Suspected Transmission of Infectious Agent by Study Drug | 0 | 0 | 0

2. Primary Outcome: Incidence of Ocular Adverse Events in the Fellow Eye
Description: This is an analysis of participants with at least one ocular adverse event (AE) that occurred in the study eye. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of the seriousness, severity, and causality for each AE. AEs of special interest (AESI) included the following: Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, are associated with severe intraocular inflammation (IOI), or require surgical or medical intervention to prevent permanent loss of sight; suspected transmission of an infectious agent by the study drug; and, cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: From the date of first administration of faricimab through 28 days after the end of study (up to 2 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Cohort A: Faricimab PTI (Prior Faricimab) | Main Study Cohort B: Faricimab PTI (Prior Aflibercept) | Substudy: Faricimab PTI
Number analyzed (Participants) | 520 | 505 | 113
Participants
  Any Adverse Event (AE), Any Severity | 157 | 149 | 17
  Serious Adverse Event (SAE) | 4 | 11 | 1
  Any AE of Special Interest (AESI) | 3 | 11 | 1
  AESI: Drop in Visual Acuity Score ≥30 Letters | 3 | 8 | 0
  AESI: Associated with Severe IOI | 0 | 0 | 0
  AESI: Intervention Required to Prevent Permanent Vision Loss | 0 | 3 | 1
  AESI: Suspected Transmission of Infectious Agent by Study Drug | 0 | 0 | 0

3. Primary Outcome: Incidence and Severity of Non-Ocular Adverse Events, With Severity Determined According to Adverse Event Severity Grading Scale
Description: This is an analysis of participants with at least one non-ocular (systemic) adverse event (AE). Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of the seriousness, severity (e.g., mild, moderate, or severe intensity), and causality for each AE. AEs of special interest (AESI) included the following: Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, are associated with severe intraocular inflammation (IOI), or require surgical or medical intervention to prevent permanent loss of sight; suspected transmission of an infectious agent by the study drug; and, cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: From the date of first administration of faricimab through 28 days after the end of study (up to 2 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Cohort A: Faricimab PTI (Prior Faricimab) | Main Study Cohort B: Faricimab PTI (Prior Aflibercept) | Substudy: Faricimab PTI
Number analyzed (Participants) | 520 | 505 | 113
Participants
  Any Adverse Event (AE), Any Severity | 343 | 337 | 41
  AE by Severity: Mild | 122 | 120 | 15
  AE by Severity: Moderate | 138 | 124 | 17
  AE by Severity: Severe | 83 | 93 | 9
  Serious Adverse Event (SAE) | 110 | 127 | 13
  AE Leading to Withdrawal from Study Treatment | 3 | 9 | 0
  Any AE of Special Interest (AESI) | 0 | 0 | 0
  AESI: Elevated ALT or AST with Either Elevated Bilirubin or Clinical Jaundice | 0 | 0 | 0

4. Primary Outcome: Substudy: Percent Change in Corneal Endothelial Cell Density From Baseline at 1 Year in the Study Eye as Compared With the Fellow Eye
Description: Specular microscopy was performed for both eyes prior to application of any topical ophthalmic anesthetic, tonometry, or any other study treatment on the same day for the evaluation of corneal endothelial cell (CEC) density. The 1-year timepoint was defined as the earliest substudy visit closest to Week 52 occurring between Week 48 and Week 64. Data (from both study eye and fellow eye) collected after the fellow eye's use of prohibited therapies-such as faricimab, brolucizumab, bevacizumab, and Port Delivery System implantation-were excluded from the corneal endothelial cell analysis.
Time Frame: Baseline and 1 year
Population: Modified Intent-to-Treat Population: All enrolled participants who received at least one injection of faricimab in the study eye during this substudy. Only participants who completed the Year 1 visit within the analysis window (Weeks 48 to 64) were included for analysis.
Measure: Mean (95% Confidence Interval); unit: Percent change in cell density
Units Other Than Participants: Eyes
Groups:
- Substudy: Faricimab PTI in the Study Eye: This analysis group represents the results for the substudy participants' study eyes. Participants from the main long-term extension study who also consented to participate in this substudy received faricimab 6 mg by intravitreal (IVT) injection into the study eye according to the personalized treatment interval (PTI) dosing regimen for the duration of the study.
- Substudy: Fellow Eye: This analysis group represents the results for the substudy participants' fellow (non-study) eyes. The participant's fellow eye was not assigned to an intervention. At the discretion of the principal investigator, a participant may have had their fellow eye treated with anti-VEGF therapy licensed for ocular use if the participant was diagnosed with an ocular condition for which the selected anti-VEGF therapy was approved by the country's regulatory agency. Administration of the following therapies to the fellow eye were prohibited during the substudy: faricimab, brolucizumab, bevacizumab, and Port Delivery System implantation.
Arm/Group | Substudy: Faricimab PTI in the Study Eye | Substudy: Fellow Eye
Number analyzed (Participants) | 99 | 99
Number analyzed (Eyes) | 99 | 99
Percent change in cell density | -0.51 [-1.68 to 0.65] | -0.71 [-1.53 to 0.10]
Statistical Analysis 1: Comparison: Substudy: Faricimab PTI in the Study Eye vs Substudy: Fellow Eye; No formal hypothesis testing was planned for this study. The paired t-tests were for reference purposes and thus not considered formal. The test was 2-sided, with the null hypothesis of no difference in percent change from baseline between the study eye and fellow eye in each patient; Test type: Other; p = 0.7702, Paired t-test; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-1.14 to 1.54] — Difference is the result of study eye minus fellow eye

5. Secondary Outcome: Substudy: Percent Change in Corneal Endothelial Cell Density From Baseline at Week 24 in the Study Eye as Compared With the Fellow Eye
Description: Specular microscopy was performed for both eyes prior to application of any topical ophthalmic anesthetic, tonometry, or any other study treatment on the same day for the evaluation of corneal endothelial cell (CEC) density. The Week 24 timepoint was defined as the earliest substudy visit closest to Week 24 occurring between Week 20 and Week 28. Data (from both study eye and fellow eye) collected after the fellow eye's use of prohibited therapies-such as faricimab, brolucizumab, bevacizumab, and Port Delivery System implantation-were excluded from the corneal endothelial cell analysis.
Time Frame: Baseline and Week 24
Population: Modified Intent-to-Treat Population: All enrolled participants who received at least one injection of faricimab in the study eye during this substudy. Only participants who completed the midpoint visit within the analysis window (Weeks 20 to 28) were included for analysis.
Measure: Mean (95% Confidence Interval); unit: Percent change in cell density
Units Other Than Participants: Eyes
Arm/Group | Substudy: Faricimab PTI in the Study Eye | Substudy: Fellow Eye
Number analyzed (Participants) | 103 | 103
Number analyzed (Eyes) | 103 | 103
Percent change in cell density | -0.02 [-0.86 to 0.81] | -0.29 [-0.92 to 0.33]
Statistical Analysis 1: Comparison: Substudy: Faricimab PTI in the Study Eye vs Substudy: Fellow Eye; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.6305, Paired t-test; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.84 to 1.38] — Difference is the result of study eye minus fellow eye

ADVERSE EVENTS:
Time Frame: From the date of first administration of faricimab through 28 days after the end of study (up to 2 years)
Description: Safety-Evaluable Population. The participants' fellow eyes were not assigned to an intervention. Ocular adverse events are included in the reported number per term, regardless of whether they occurred in the study eye or the fellow eye.
Arm/Group | Main Study Cohort A: Faricimab PTI (Prior Faricimab) | Main Study Cohort B: Faricimab PTI (Prior Aflibercept) | Substudy: Faricimab PTI
All-Cause Mortality (participants affected / at risk) | 13/520 | 27/505 | 1/113
Serious Adverse Events (participants affected / at risk) | 125/520 | 156/505 | 14/113
Other Adverse Events (participants affected / at risk) | 158/520 | 169/505 | 9/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Cohort A: Faricimab PTI (Prior Faricimab) (N=520) | Main Study Cohort B: Faricimab PTI (Prior Aflibercept) (N=505) | Substudy: Faricimab PTI (N=113)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 4 (4) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (2) | 1 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 5 (5) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 6 (6) | 7 (7) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 6 (6) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Age-related macular degeneration (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 5 (5) | 7 (7) | 0 (0)
Choroidal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 4 (4) | 14 (14) | 0 (0)
Non-infectious endophthalmitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Retinal aneurysm (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2) | 1 (2)
Retinal pigment epithelial tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Subretinal fibrosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 3 (3) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenogastric reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (3) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 3 (3) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Physical deconditioning (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 5 (5) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dermo-hypodermitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 9 (9) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4) | 1 (1)
Viral uveitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Failed back surgery syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 7 (7) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Shoulder fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stoma obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0)
Inflammatory marker increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Starvation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ameloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Eyelid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Urethral cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 5 (6) | 1 (1)
Cognitive disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Drop attacks (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Device loosening (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depressive delusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (4) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephritic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatic disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Cohort A: Faricimab PTI (Prior Faricimab) (N=520) | Main Study Cohort B: Faricimab PTI (Prior Aflibercept) (N=505) | Substudy: Faricimab PTI (N=113)
Cataract (Eye disorders) | 56 (78) | 63 (80) | 2 (2)
Neovascular age-related macular degeneration (Eye disorders) | 60 (70) | 55 (65) | 2 (3)
Posterior capsule opacification (Eye disorders) | 14 (17) | 26 (30) | 1 (1)
COVID-19 (Infections and infestations) | 61 (65) | 48 (49) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (4):
  • Study Protocol: Main Study (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT04777201/Prot_000.pdf
  • Study Protocol: CEC Substudy (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT04777201/Prot_001.pdf
  • Statistical Analysis Plan: Main Study (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT04777201/SAP_002.pdf
  • Statistical Analysis Plan: CEC Substudy (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT04777201/SAP_003.pdf